CLINICAL TRIAL: NCT05814549
Title: A Study of Using Plasma Circulating Cell Free Human Papillomavirus Deoxyribonucleic Acid to Screen (cf HPV DNA) for HPV-Related Oropharyngeal Cancer
Brief Title: A Study Using Human Papillomavirus (HPV) DNA Testing to Detect HPV-Related Oropharyngeal Cancer (OPC)
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 22-234
Record Dates: First submitted 2023-04-03; First posted 2023-04-18 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Oropharyngeal Cancer; HPV-Related Carcinoma; HPV Positive Oropharyngeal Squamous Cell Carcinoma
Keywords: HPV-Related Oropharyngeal Cancer; Human Papillomavirus; Oropharyngeal Cancer; HPV-Related Carcinoma; HPV Positive Oropharyngeal Squamous Cell Carcinoma; Cell Free Human Papillomavirus Deoxyribonucleic Acid; cf HPV DNA; 22-234; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Oropharyngeal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No previous history of diagnosed HPV-related head and neck cancer: Participants have no previous history of diagnosed HPV-related head and neck cancer
  Interventions: Diagnostic Test: NavDx

INTERVENTIONS:
Diagnostic Test: NavDx — Evaluation of HPV presence via NavDx (v1) at two (or three) timepoints
  o If one of the two blood samples is positive, the subject will have a third NavDx (v1) test approximately 1 month after the second timepoint. If the test is positive, the subject will move to surveillance phase.

SUMMARY:
The researchers think that a blood test (NavDx®) may be able to identify cancer early by looking for circulating DNA from Human Papillomavirus/HPV. Circulating DNA are small pieces of genes that are released into the bloodstream. The purpose of this study is to find out whether using this blood test to test for HPV DNA will help detect HPV-related Oropharyngeal Cancer/OPC.

ELIGIBILITY:
Inclusion Criteria:

* Ages 45 and older
* Self-reported history of four or more lifetime sexual partners
* Self-reported history of one or more lifetime oral sexual partner
* No previous history of diagnosed HPV-related head and neck cancer

Exclusion Criteria:

* History of diagnosed HPV-related OPC
* Less than three sexual partners in lifetime
* No history of oral sex performed
* Younger than age 45

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential research participants will be identified by a member of the patient's treatment team, the protocol investigator, or research team at Memorial Sloan-Kettering Cancer Center (MSKCC). If the investigator is a member of the treatment team, s/he will screen their participant's medical records for suitable research study participants and discuss the study and their potential for enrolling in the research study. Potential participants contacted by their treating physician will be referred to the investigator/research staff of the study
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2031-03-31 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants found to have HPV-related OPC | Up to 5 years
  : The primary objective is to determine the feasibility of screening by estimating the yield (proportion of subjects found to have HPV-related OPC out of all subjects screened).

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Lee, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk- Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org